CLINICAL TRIAL: NCT00111488
Title: Randomized Study of Surgical Ablation With Microwave Energy for the Treatment of Atrial Fibrillation
Brief Title: Guidant Microwave Ablation System for the Treatment of Atrial Fibrillation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: VR2045885
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2014-05

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radionuclide Generators

INTERVENTIONS:
Device: Flex 4 and Generator

SUMMARY:
The purpose of the Randomized Study of Surgical Ablation with Microwave Energy for the Treatment of Atrial Fibrillation (RESOLVE-AF) trial is to determine the safety and effectiveness of the Guidant FLEX® Microwave Surgical Ablation System in the treatment of permanent atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

* Patient age >= 18 years
* Documented permanent AF (for at least three months)
* Scheduled for an open chest cardiac surgery for the primary indication of mitral valve repair or replacement
* Has been informed of the nature of the study, agrees to its provisions, and provided written informed consent, which was approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site

Exclusion Criteria:

* Cerebral vascular accident (CVA, stroke) or transient ischemic attack (TIA) within the previous 6 months
* Myocardial infarction within the previous 6 weeks
* Documented history of pulmonary vein stenosis
* Previous ablation attempt for AF
* Previous thoracic procedures
* Left atrial size > 7.0 cm
* Left ventricular ejection fraction < 30%
* Presence of left atrial or left atrial appendage thrombi
* Esophageal fistula or other stricture, untreated esophagitis, varices, dysphagia or odynophagia contraindicating transesophageal echocardiography
* Known allergy or contraindication to warfarin therapy
* Known allergy or contraindication to antiarrhythmic (Classes IA, IC, III) therapy
* Other comorbidity with reduced life expectancy of less than 1 year or protocol noncompliance that would limit follow-up
* Geographically remote or unable to return for follow-up examinations
* Pregnant or planning to become pregnant during the study
* Enrolled in any concurrent study, without Guidant written approval, that may confound the results of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial fibrillation at six months
Composite major adverse event at one month | One month

SECONDARY OUTCOMES:
Composite Majour Adverse Events at three and 6 months | 3 months and 6 months
Restoration of normal sinus rhythm at discharge | Hospital discharge
Change in cardiac function at six month | 6 month
Change in Quality of Life at six months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mack, MD, Principal Investigator — Cardiopulmonary Research Science and Technology Institute
Locations (21):
- United States (21):
  - Scripps Memorial/ Kaiser Permanente, La Jolla, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Mercy General Hospital, Sacramento, California
  - Piedmont Hospital, Atlanta, Georgia
  - Methodist Hospital, Indianapolis, Indiana
  - St. Francis Hospital and Health Center, Indianapolis, Indiana
  - Alegent Health, Omaha, Nebraska
  - St. Michael's Medical Center, Newark, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Lenox Hill Hospital, New York, New York
  - Univesity of Rochester Medical, Rochester, New York
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cardiopulmonary Research Science and Technology Institute, Dallas, Texas
  - Baylor University, Dallas, Texas
  - Plaza Medical Center, Fort Worth, Texas
  - University of VIrginia Health System, Charlottesville, Virginia
  - Virginia Masonic Clinic, Seattle, Washington
  - Wisconsin Heart Hospital, Milwaukee, Wisconsin
  - Wausau Heart and Lung Surgeons, Wausau, Wisconsin